CLINICAL TRIAL: NCT04832776
Title: FOLFOXIRI Plus Cetuximab Versus FOLFOXIRI Plus Bevacizumab in Conversion Therapy of Right-sided Colon Cancer Liver Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Sanjun Cai, Department of Colorectal Surgery, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cetu-Bev-FOLFOXIRI
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Liver Metastasis Colon Cancer
Keywords: FOLFOXIRI; cetuximab; bevacizumab
MeSH Terms: interventions — Cetuximab; Bevacizumab; FOLFOXIRI protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FOLFOXIRI+C225 (Experimental)
  Interventions: Drug: Cetuximab; Drug: FOLFOXIRI
- FOLFOXIRI+BEV (Active Comparator)
  Interventions: Drug: Bevacizumab; Drug: FOLFOXIRI

INTERVENTIONS:
Drug: Cetuximab — one group plus cetuximab
  Arms: FOLFOXIRI+C225
Drug: Bevacizumab — one group plus bevacizumab
  Arms: FOLFOXIRI+BEV
Drug: FOLFOXIRI — FOLFOXIRI

SUMMARY:
To compare the efficacy of FOLFOXIRI plus Cetuximab and FOLFOXIRI plus Bevacuzumab in the conversion therapy of right-sided colon cancer liver metastases

ELIGIBILITY:
Inclusion Criteria:

* ECOG perfomance 0-1
* pathologically confirmed colorectal carcinoma, with RAS wild type
* inital unresectable liver metastases discussed by MDT
* prior no systemical therapy or exceed 6 months after the adjuvant chemotherapy of primary tumor surgery.
* without extraheptic metastatic lesions, except for locally controlled lung metastases (RFA or SBRT)
* adequate blood, liver and renal function
* expected survival longer than 6 months

Exclusion Criteria:

* with bleeding risk
* interestinal obstruction or disease
* uncontrolled hypertension and severe heart disease
* previous severe thrombotic events
* central nervous system metastases
* accompanied with other malignant tumor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-04-17 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 8 weeks
  objective response rate

SECONDARY OUTCOMES:
R0 resection rate of liver metastases | up to 8 weeks
  R0 resection rate of liver metastases
NED rate | up to 8 weeks
  percentage of patients who reach NED
OS | up to 6 months
  overal survival
PFS | up to 8 weeks
  progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Wen Zhang, Principal Investigator — Fudan University
Locations (1):
- Department of Colorectal Surgery Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China